CLINICAL TRIAL: NCT02249897
Title: PRELIMINARY EVALUATION OF RETINAL EFFECTS OF PHARMACOLOLOGICAL LOWERING OF SERUM LEVES OF ADVANCED GLYCATION END-PRODUCTS (AGEs) IN TYPE 2 DIABETIC PATIENTS
Brief Title: PRELIMINARY EVALUATION OF PHARMACOLOGICAL LOWERING OF AGEs
Acronym: PREL-AGES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Clinica Alemana de Santiago (Other)
Responsible Party: Principal Investigator, MARIA PIA DE LA MAZA, Professor, University of Chile
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: AGE-1
Record Dates: First submitted 2014-09-17; First posted 2014-09-26 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: DIABETES; DIABETIC RETINOPATHY; DIABETIC NEUROPATHY
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy; Diabetic Neuropathies | interventions — Cholestyramine Resin

STUDY DESIGN:
Intervention Model Description: Prescription of 6 g oral cholestiramine in 7 patients with type 2 DM, to study changes in neuroophtalmologic variables (electroretinogram and optic nerve conduction)
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PLACEBO (Placebo Comparator): AFTER COMPLETING THE INITIAL EVALUATION (ANTHROPOMETRY, SERUM BIOCHEMISTRY AND CML LEVELS, FUNDUS, MUTIFOCAL ELECTRORETINOGRAM AND OPTIC NERVE CONDUCTION VELOCITY) PATIENTS WILL RECEIVE ORAL PLACEBO CAPSULES 4 PER EACH MEAL/DAY DURING 12 WEEKS
  Interventions: Drug: CHOLESTYRAMINE
- CHOLESTIRAMINE (Active Comparator): AFTER COMPLETING THE CONTROL PERIOD (PLACEBO CAPSULES) PATIENTS WILL BE REASSESSED, AND THEN TREATED WITH ORAL CHOLESTYRAMINE 6 G/DAY (500 MG CAPSULES -> 4 CAPSULES PER EACH MEAL/DAY) DURING 12 WEEKS AND E SAME INITIAL EVALUATION WILL BE REPEATED
  Interventions: Drug: CHOLESTYRAMINE

INTERVENTIONS:
Drug: CHOLESTYRAMINE — CHOLESTYRAMINE CAPSULES, 6 G/DAY P.O. DURING 12 WEEKS
  Other Names: QUESTRAN

SUMMARY:
There is evidence of the association between diabetic microangiopathy and elevated serum concentrations of advanced glycation end-products (AGEs). AGEs levels are associated with ingestion of specific foods (baked meats and milk powder); reducing their dietary intake lowers AGEs concentrations, with beneficial metabolic effects; however threre is still no evidence of whether this has an impact on microvascular complications of DM. We recently applied for funding to compare in a RCT the effects of Cholestyramine versus placebo, on visual electrophysiology. This drug is similar to Sevelamer in structure, both act as chelators of bile salts, and reduce absorption of dietary AGE, lowering serum levels. However it is essential to carry out preliminary tests to assess aspects that may imply adjustments to the proposed protocol, such as: 1) tolerance to the drug 2) short term effect of the drug versus placebo on serum levels of AGEs 3) effects of the drug versus placebo in levels of fat soluble vitamins (D and K specifically) 4) intra and interindividual variability of electrophysiological measurements of vision (ERGMF and optic nerve conduction velocity) 5) drug versus placebo in electrophysiological measurements of vision (neuroconduction ERGMF and optic nerve). Objective: The present project is planned as a pilot study, which will clarify points 1 to 5. Methodology: patients (6 DM2, 25 -50 y) will be assessed through anthropometry, clinical laboratory tests (creatinine, chemistry profile, lipid profile, microalbuminuria glycosylated hemoglobin, vitamin B12, 25OH vitamin D and prothrombin), dietary recalls specifically designed to analyze the regular consumption of AGEs, serum CML and neuro-ophthalmological study (fundus, ERGMF and optic nerve conduction). Subsequently each patient will be assigned to treatment with placebo for 3 months and then Cholestyramine 6 g / day for 12 weeks and at the end of each period will be reassessed using the same methodology. If patients cannot tolerate the drug, they will be assigned to a reduced AGE diet.

Expected results: Cholestyramine will have side effect similar to placebo (mainly digestive). The active drug and not placebo will reduce serum levels of AGEs and electrophysiological parameters of vision at 12 weeks. It is expected that a low AGEs diet in patients who do not tolerate the drug will also reduce serum CML although to a lesser degree and will also induce electrophysiologic changes.

DETAILED DESCRIPTION:
Patients: 6 adults with type 2diabetes will be selected, ages between 25 and 50 years, with more than 5 and less than 10 years of disease, adherent to treatment with oral hypoglycemic agents or insulin, who agree to participate in the study through a written informed consent. Only those with a high habitual intake of AGEs according the food recall will be included. Patients with the following characteristics will be excluded: -Severe Obesity (BMI> 35 kg / m2), glycosylated hemoglobin> 9%, anemia, renal failure (creatinine> 1.5 mg / dL or calculated creatinine clearance <60 ml / min), fasting plasma glucose> 250 mg / dL or a history of acute hyperglycemic complications requiring hospitalization in the past 2 years, severe diabetic dyslipidemia (LDL> 130, TG> 350 mg / dL) or vitamin B12 deficiency, a history of heart, liver, lung cancer or chronic diseases, clinical diagnosis of diabetic neuropathy and eye conditions that could hinder electroretinogram, such as uncorrected refractive defects, cataracts and severe diabetic retinopathy or macular edema. Other exclusion criteria will be poorly controlled hypertension or acute vascular event in the past 2 years and pregnancy.

After signing an informed consent, patients will undergo the following assessments: 1) History and drug registration. 2) dietary survey including methods of food preparation, consumption of dietary products containing fructose or corn starches and specific foods rich in AGEs according to measurements made in Chilean foods (milk and concentrated powder, biscuits, cheeses was also specifically recorded, roasted meats and grilled sausages etc.). 3) anthropometry (weight, height, waist circumference) 4) fasting basic laboratory tests fasting (hemoglobin, TSH, glucose, glycosylated hemoglobin, creatinine, prothrombin, lipid profile and serum levels of vitamin B12 and vitamin D), using automated clinical laboratory techniques. 5) morning urine for determination of microalbuminuria (MAU / creatinine) 6) Inflammatory markers (ultrasensitive PCR) using a commercial ELISA kit. 7) Concentration of serum AGEs (CML through Abcam ELISA Antibody) 8) Visual evoked potentials as indicator of electrophysiological conduction after visual stimulation through the optic nerve (ON) exploring the visual pathway (myelin) to the occipital cortex. 9) ophtalmologic examination with biomicroscopy for evaluation of refractive defects and fundus (to diagnose the presence or absence of retinopathy) and evoked potentials by multifocal electroretinography.

This series of evaluations will be repeated after each each treatment period of 12 weeks each, ie on 3 occasions. Indications and reinforcement of traditional dietary measures to improve glycemic control (restriction of caloric intake according to body composition, decrease of intake of simple carbohydrates and increase of soluble and insoluble fiber to reduce glycemic load), according to the standards for diabetes management from the Ministry of Health. Also if necessary the hypoglycemic or insulin therapy will be adjusted in order to achieve adequate metabolic control (HbA1c <7%).

For the specific drug treatment, initially inert placebo (talc) capsuleswill be prescribed during 12 weeks then switching to Cholestyramine during 12 weeks, with equal physical characteristics of capsules, after which all initial evaluations be repeated. Cholestyramine treatment will be prescribed using a 6 g daily dose (4 tablets daily of 500 mg each of cholestyramine with each main meal). Patients that manifest adverse effects with the use of the active drug and cannot maintain the treatment, will be assigned to a dietary treatment with a reduced AGE diet according to the recommendations of Uribarri et. al. (32) for 12 weeks, at the end of which the initial evaluation will be repeated. In both periods supplementation with vitamin D in doses adjusted to pre-intervention, vitamin A and E in adequate doses to meet the DRI level and vitamin K if needed will be prescribed. Patients will be monitored monthly by their treating diabetologist, verifying compliance, registering adverse events, anthropometric measurements and fasting blood glucose. If elevated blood glucose levels are detected infectious causes or failure to adhere dietary indications will be discarded and corrective measures will be initiated. In patients who do not meet the inclusion criteria due to vitamin B12 deficiency, intramuscular supplementation will be indicated and will be referred to their respective centers. If vitamin D deficiency is detected, proper supplementation before entering the study will be indicated. At the end of the control period (placebo for 12 weeks), the same initial assessments will be repeated and then a second treatment (cholestyramine 6 g / day) will be assigned, repeating the same assessments at the end of these 3 months.

Blood samples for determination of CML and ultrasensitive PCR will remain frozen at -70 degrees to be processed all at the end of the study, avoiding to make any technical changes on 2 times. Instead determinations to be made in clinical laboratory (TSH, prothrombin, glycemia, lipid profile, creatinine, glycated hemoglobin, microalbuminuria and levels of vitamins B12 and D), will be processed immediately, delivering a copy of the results to each patient to facilitate corrective measures necessary.

Primary endpoint and sample size: For this pilot study sample size was not estimated because one of the objectives is to assess variability and detect whether the short period of treatment does induce changes in electrophysiological variables that are clearly detectable, in addition to assessing drug tolerance. With this information you can better estimate the sample size for a randomized controlled larger. In addition it was felt necessary to begin the study using the placebo and no treatment assigned randomly because washout period would be necessary for a randomized crossover study of random type is unknown. The proposed (6 patients) sample size was calculated based on the available budget. It is important to note that analysis of evoked potentials and electroretinography considers each eye separately, so that there will be 12 eyes in 6 patients.

ELIGIBILITY:
Inclusion Criteria:

* TYPE 2 DIABETES
* More than 5 and less than 10 years of disease
* Adherent to treatment with oral hypoglycemic agents or insulin
* Agree to participate in the study through a written informed consent.
* High habitual intake of AGEs according the food recall .

Exclusion Criteria:

* Severe Obesity (BMI> 35 kg / m2)
* Glycosylated hemoglobin> 9%, anemia, renal failure (creatinine> 1.5 mg / dL or calculated creatinine clearance <60 ml / min), fasting plasma glucose> 250 mg / dL
* History of acute hyperglycemic complications requiring hospitalization in the past 2 years
* Severe diabetic dyslipidemia (LDL> 130, TG> 350 mg / dL)
* Vitamin B12 deficiency
* History of heart, liver, lung cancer or chronic diseases
* Clinical diagnosis of diabetic neiropathy and eye conditions that could hinder electroretinogram, such as uncorrected refractive defects, cataracts and severe diabetic retinopathy or macular edema.
* Poorly controlled hypertension or acute vascular event in the past 2 years
* Pregnancy.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
CML SERUM LEVELS | 12 WEEKS
  REDUCTION OF CARBOXYMETHYL (CML) SERUM LEVELS

SECONDARY OUTCOMES:
OPTICAL NERVE CONDUCTION | 12 WEEKS
  CHANGE IN OPTICAL NERVE CONDUCTION AFTER VISUAL STIMULUS RESPECT PLACEBO
MULTIFOCAL ELECTRORETINOGRAPHY | 12 WEEKS
  SIGNIFICANT CHANGE RESPECT PLACEBO

CONTACTS AND LOCATIONS:
Overall Officials: MARIA PIA DE LA MAZA, PROFESSOR, Principal Investigator — INSTITUTE OF NUTRITION & FOOD TECHNOLOGY, UNIVERSITY OF CHILE
Locations (2):
- Chile (2):
  - Institute of Nutrition & Food Technology (INTA), Santiago, Metropolitan Region
  - Clinica Alemana de Santiago, Santiago, Santiago Metropolitan